CLINICAL TRIAL: NCT01748903
Title: TARGET Intracranial Aneurysm Coiling Registry: A Prospective Clinical Efficacy and Safety Study of Stryker Target® 360°, Target® Helical, and 2nd Generation Target® Nano Coils
Brief Title: TARGET Intracranial Aneurysm Coiling Registry
Acronym: TARGET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mercy Health Ohio (Other)
Collaborators: Stryker Neurovascular (Industry)
Responsible Party: Principal Investigator, Dr. Osama O. Zaidat, Medical Director, Neuroscience and Stroke Programs, Mercy Health Ohio
Other Study IDs: 19180
Record Dates: First submitted 2012-12-07; First posted 2012-12-13 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Intracranial Aneurysms
Keywords: intracranial aneurysm; cerebral aneurysm; packing density; Target Coils; aneurysm embolization
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Target 360°, 2D, Nano Coils: Subjects will undergo embolization using Target 360°, 2D, Nano Coils for the treatment of their intracranial aneurysm.
  Interventions: Device: Target 360°, 2D Coils, Nano Coils

INTERVENTIONS:
Device: Target 360°, 2D Coils, Nano Coils
  Other Names: Target coils; Target Nano coil

SUMMARY:
The purpose of this prospective registry is to collect real world, post-marketing data on the use of Stryker Target® 360,Target® 2D, and 2nd generation Target® Nano coils for the embolization of ruptured or unruptured intracranial saccular aneurysms. Up to 300 patients (150 in the TARGET 360°/Helical arm and 150 in the New NANO arm) presenting with intracranial aneurysms suitable for coil embolization will be enrolled at up to 20 sites. A post hoc analysis comparing Target® 360° and Target® 2D coil technical and clinical endpoints will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 18 years or older.
2. Patient has a documented, previously untreated, saccular intracranial aneurysm, unruptured or ruptured, suitable for embolization with coils.
3. (NEW NANO arm ONLY) Target aneurysm is ≤7mm.
4. Patient has a Hunt and Hess Score of 3 or less.
5. Patient has a premorbid mRS of 3 or less.
6. Patient or patient's legally authorized representative has provided written informed consent.
7. Patient is willing to and can comply with study follow-up requirements.

Exclusion Criteria:

1. Patient is < 18 years old.
2. Dissecting aneurysm.
3. Patients with intracranial aneurysms (other than the target aneurysm) that will require treatment during the study period (enrollment through follow-up).
4. Patients in whom the target aneurysm will be treated with coils other than Stryker Target® 360°, Target® Helical coils, and 2nd generation Target® Nano Coils.
5. (NEW NANO Arm ONLY) Patients in whom the target aneurysm was treated with a total coil length comprised of <25% Stryker Target® 2nd generation Nano Coils.
6. Target aneurysm is fusiform.
7. Patients in which the target aneurysm cannot be coiled in one procedure (i.e. staged procedure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All sequential patients presenting with unruptured and ruptured saccular aneurysms, who meet all eligibility criteria, will be considered for study enrollment.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-02; Primary Completion 2019-01 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Packing Density | At immediate post-procedure (Day 1)
  Packing density will be calculated based on aneurysm volume and amount of coil used during the embolization procedure.

SECONDARY OUTCOMES:
Occlusion Rate | At immediate post-procedure (Day 1) and 3-9 month follow-up
  Angiographic occlusion of the aneurysm will be adjudicated by an independent core lab using immediate post-procedure and 3-9 month follow-up angiography.
Aneurysm Re-access Rate | At end of study procedure (Day 1)
  The rate of re-assess (Microcatheter kick-back rate) of the target aneurysm will be captured during the procedure.
Time of Fluoroscopic Exposure | At immediate post-procedure (Day 1)
  Total time of fluoroscopic exposure will be captured from the initial recording of the road map to the final angiogram after completion of the coil embolization procedure.
Overall Procedure Time | At Immediate post-procedure (Day 1)
  The overall procedure time will be captured from the time of guide catheter placement to the end of the coil embolization procedure.
Aneurysm Recurrence | 3-9 month follow-up
Aneurysm Re-treatment Rate | 3-9 month follow-up
  Aneurysm re-treatment rates will be tracked and recorded during the 3-9 month follow-up
Aneurysm Bleed and Re-bleed Rate | 3-9 month follow-up
  Aneurysm Bleed and Re-bleed Rate will be assessed and recorded at the 3-9 month follow-up.
Treatment-related Morbidity and Mortality | from study procedure (Day 1) to 3-9 month follow-up
  Treatment-related morbidity and morality will be tracked and recorded from study procedure through the 3-9 month follow-up.
Modified Rankin Score | At baseline (Day 1) and hospital discharge (Day 3) and 3-9 month follow-up
  Modified Rankin score will be recorded at baseline, hospital discharge, and during the 3-9 month follow-up.
Device-related serious adverse events | From the study procedure (Day 1) until 3-9 month follow up
  Procedural and post-procedural serious adverse events related to the device and/or procedure will be captured and recorded at the end of the procedure and until the patient has completed the 3-9 month follow-up.
Length of hospital stay | At hospital discharge (Day 3)
  Length of hospital stay will be recorded at the time of patient discharge.
Technical and clinical endpoints of Target 360° and 2D coils | 3-9 month follow-up
  A post hoc analysis comparing Target 360° and 2D coil primary and secondary technical and clinical endpoints will be performed upon final data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Osama O Zaidat, MD, MS, Principal Investigator — Mercy Health St. Vincent Medical Center
Locations (9):
- United States (9):
  - University of Arizona, Phoenix, Arizona
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Presence Saint Joseph Medical Center, Joliet, Illinois
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - McLaren Health, Flint, Michigan
  - SSM DePaul Health Center, St Louis, Missouri
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - Greenville Health System, Greenville, South Carolina
  - West Virginia University Hospital, Morgantown, West Virginia

REFERENCES:
- [Derived] Zaidat OO, Castonguay AC, Rai AT, Badruddin A, Mack WJ, Alshekhlee AK, Shah QA, Hussain SI, Kabbani MR, Bulsara KR, Taqi AM, Janardhan V, Patterson MS, Nordhaus BL, Elijovich L, Puri AS. TARGET(R) Intracranial Aneurysm Coiling Prospective Multicenter Registry: Final Analysis of Peri-Procedural and Long-Term Safety and Efficacy Results. Front Neurol. 2019 Jul 9;10:737. doi: 10.3389/fneur.2019.00737. eCollection 2019. PMID 31338061